CLINICAL TRIAL: NCT06058793
Title: Brightline-4: A Phase III Open-label, Single-arm, Multi-center Study to Assess the Safety and Efficacy of Brigimadlin (BI 907828) Treatment in Patients With Treatment-naïve or Pre-treated Advanced Dedifferentiated Liposarcoma
Brief Title: Brightline-4: A Study to Test How Well Brigimadlin is Tolerated by People With a Type of Cancer Called Dedifferentiated Liposarcoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1403-0019; 2023-504522-19-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2023-09-22; First posted 2023-09-28 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Liposarcoma, Dedifferentiated
MeSH Terms: conditions — Liposarcoma | interventions — brigimadlin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Brigimadlin treatment (Experimental)
  Interventions: Drug: Brigimadlin

INTERVENTIONS:
Drug: Brigimadlin — Brigimadlin
  Other Names: BI 907828

SUMMARY:
This study is open to adults with a type of cancer called dedifferentiated liposarcoma (DDLPS). They can join the study if their tumours are positive for MDM2. The purpose of this study is to find out whether a medicine called brigimadlin (BI 907828) is tolerated by and helps people with DDLPS. Brigimadlin is a so-called MDM2 inhibitor that is being developed to treat cancer.

Participants take brigimadlin as a tablet once every 3 weeks. Participants may continue to take brigimadlin as long as they benefit from treatment and can tolerate it. They visit the study site regularly. At the study site, doctors regularly check participants' health and take note of any unwanted effects. The doctors also regularly check tumour size.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent form (ICF) in accordance with International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH) - Good Clinical Practice (GCP) and local legislation prior to any study-specific procedures, sampling, or analyses
2. Male or female patients ≥18 years old at the time of signature of the ICF
3. Women of childbearing potential (WOCBP) and men able to father a child must be ready and able to use two medically acceptable methods of birth control per ICH M3 (R2) that result in a low failure rate of <1% per year when used consistently and correctly beginning at screening, during study participation, and until 6 months and 12 days after last dose for women and 102 days after last dose for men. A list of contraception methods meeting these criteria is provided in the patient information
4. Histologically documented locally advanced or metastatic, unresectable (i.e. surgery morbidity would outweigh potential benefits), progressive or recurrent Dedifferentiated liposarcoma (DDLPS), meeting the criteria for an open study cohort:

   * Cohort A: patient has not received prior systemic therapy for DDLPS in any setting (including adjuvant, neoadjuvant, maintenance, palliative)
   * Cohort B: patient has received any prior systemic therapy for DDLPS in any setting (including adjuvant, neoadjuvant, maintenance, palliative)
5. Written pathology report indicating the diagnosis of DDLPS with positive MDM2 immunohistochemistry or MDM2 amplification as demonstrated by fluorescence in situ hybridisation (FISH) or next-generation sequencing (NGS)
6. Presence of at least 1 measurable target lesion according to RECIST version 1.1. In patients who only have 1 target lesion, the baseline imaging must be performed at least 2 weeks after any biopsy of the target lesion
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
8. Life expectancy ≥3 months at the start of treatment in the opinion of the investigator Further inclusion criteria apply.

Exclusion Criteria:

1. Known mutation in the TP53 gene (screening for TP53 status is not required)
2. Major surgery (major according to the investigator's assessment) performed within 4 weeks prior to start of study treatment or planned within 6 months after screening
3. Previous administration of brigimadlin or any other MDM2-p53 or MDM4 regulator of p53 (MDM4/MDMX)-p53 antagonist
4. Previous treatment in study 1403-0008 (Brightline-1)
5. Having to receive, or intending to receive, restricted medications or any drug considered likely to interfere with the safe conduct of the study
6. Receiving treatment for brain metastases or leptomeningeal disease (LMD) which may interfere with safety and/or endpoint assessment
7. Unable to swallow the study treatment
8. Previous or concomitant malignancies other than the one treated in this study within the previous 2 years, except effectively treated non-melanoma skin cancers, carcinoma in situ of the cervix, ductal carcinoma in situ, or other malignancy that is considered cured by local treatment Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2023-12-13 (Actual); Primary Completion 2025-12-12 (Actual); Study Completion 2025-12-12 (Actual)

PRIMARY OUTCOMES:
Occurrence of Treatment-emergent adverse events (TEAEs) according to Common Terminology Criteria for Adverse Events (CTCAE) version 5 during the entire treatment period | up to 23 months
Occurrence of TEAEs with Grade ≥3 according to CTCAE version 5 during the entire treatment period | up to 23 months

SECONDARY OUTCOMES:
Occurrence of treatment-emergent serious adverse events (SAEs) | up to 23 months
Occurrence of TEAEs leading to study treatment discontinuation | up to 23 months
Occurrence of TEAEs leading to dose reduction | up to 23 months
Occurrence of TEAEs leading to dose delay | up to 23 months
Occurrence of TEAEs of special interest (adverse events of special interest [AESIs]) | up to 23 months
Objective response (OR) | up to 23 months
  OR is defined as a best overall response of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1 (based on investigator assessment) from the date of treatment start until the earliest date of disease progression, death, last evaluable tumour assessment before start of subsequent anticancer therapy, lost to follow-up, withdrawal of consent or end of study (EoS)
Progression-free survival (PFS) | up to 23 months
  PFS is defined as the time from treatment start until the earliest date of tumour progression according to RECIST version 1.1, based on investigator assessment, or death from any cause
Overall survival (OS) | up to 23 months
  OS is defined as the time from treatment start until death from any cause
Duration of objective response (DOR) | up to 23 months
  DOR is defined as the time from first documented confirmed OR until the earliest date of disease progression or death among patients with confirmed OR (based on investigator assessment)
Disease control (DC) | up to 23 months
  DC is defined as a best overall response of CR, PR, or stable disease (SD) where best overall response is defined according to RECIST version 1.1 based on investigator assessment

CONTACTS AND LOCATIONS:
Locations (56):
- United States (26):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic-Arizona, Phoenix, Arizona
  - Precision NextGen Oncology, Beverly Hills, California
  - Sarcoma Oncology Center, Santa Monica, California
  - University of California Los Angeles, Santa Monica, California
  - Yale Cancer Center, New Haven, Connecticut
  - Mayo Clinic - Florida, Jacksonville, Florida
  - University Cancer and Blood Center, Athens, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Kansas Cancer Center, Overland Park, Kansas
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - John Theurer Cancer Center, Hackensack, New Jersey
  - Northwell Health, Lake Success, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Abramson Cancer Center at Pennsylvania Hospital, Philadelphia, Pennsylvania
  - West Cancer Center & Research Institute, Germantown, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Utah Cancer Specialists Cancer Center, Salt Lake City, Utah
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Medical Oncology Associates, P.S., Spokane, Washington
  - Froedtert and The Medical College of Wisconsin, Milwaukee, Wisconsin
- Argentina (4):
  - Hospital Britanico de Buenos Aires, CABA
  - Sanatorio Finochietto, CABA
  - Hospital Italiano de Buenos Aires, CABA
  - Instituto Medico Especializado Alexander Fleming, Ciudad Autonoma de Bs As
- Australia (4):
  - Prince of Wales Hospital-Randwick-66496, Randwick, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Brazil (5):
  - Pronutrir, Fortaleza
  - Hospital do Cancer de Londrina, Londrina
  - CEPHO - Centro de Estudos e Pesquisas em Hematologia e Oncologia, Santo André
  - Hospital Sao Domingos, São Luís
  - H.S.J. Beneficência Portuguesa - São Paulo, São Paulo
- Canada (3):
  - Arthur J. E. Child Comprehensive Cancer Centre, Calgary, Alberta
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - McGill University Health Centre (MUHC), Montreal, Quebec
- Japan (10):
  - Aichi Cancer Center Hospital, Aichi, Nagoya
  - Nagoya University Hospital, Aichi, Nagoya
  - National Cancer Center Hospital East, Chiba, Kashiwa
  - National Hospital Organization Kyushu Cancer Center, Fukuoka, Fukuoka
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Tohoku University Hospital, Miyagi, Sendai
  - Okayama University Hospital, Okayama, Okayama
  - Osaka International Cancer Institute, Osaka, Osaka
  - Hokkaido Cancer Center, Sapporo, Hokkaido
  - Japanese Foundation for Cancer Research, Tokyo, Koto-ku
- United Kingdom (4):
  - Addenbrooke's Hospital, Cambridge
  - Beatson West of Scotland Cancer Centre, Glasgow
  - The Royal Marsden Hospital, Chelsea, London
  - The Christie, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After structured results have been posted, all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com